CLINICAL TRIAL: NCT01797796
Title: A Double Blind, Randomized, Placebo-Controlled, Third-Party Open, Cross-Over Study To Examine The Effect Of PF-06305591 On Capsaicin And Capsaicin/Heat-Induced Neurogenic Flare In Healthy Volunteers
Brief Title: Effect Of PF-06305591 On Capsaicin And Capsaicin/Heat-Induced Neurogenic Flare
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5281005
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-06305591 (Experimental)
  Interventions: Drug: PF-06305591; Other: Capsaicin challenge
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Other: Capsaicin challenge

INTERVENTIONS:
Drug: PF-06305591 — 150 mg PF 06305591 will be administered to subjects as a 100 mL extemporaneous prepared oral solution once.
  Arms: PF-06305591
Other: Capsaicin challenge — 110 mg capsaicin cream (Axsain®) will be applied topically at each visit.
  Arms: PF-06305591
Drug: Placebo — Placebo will be administered to subjects as a 100 mL extemporaneous prepared oral solution once.
  Arms: Placebo
Other: Capsaicin challenge — 110 mg capsaicin cream (Axsain®) will be applied topically at each visit.
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of PF-06305591 on capsaicin and capsaicin/heat-induced neurogenic flare.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Caucasian subjects with skin type I-III inclusive (Fitzpatrick Scale), between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* An informed consent document signed and dated by the subject.
* Subjects must have a distance from base of scaphoid to antecubital fossa equal of greater to 26 cm on their forearms.
* Subjects who demonstrate a capsaicin -mediated neurogenic flare with a value >200 on the arbitrary Laser Doppler output at any of the time points 30, 40, 50 or 60 minutes following administration of capsaicin at Screening.

Exclusion Criteria:

* Evidence or history of clinically significant hematological (ie, abnormalities due to prolonged exposure to altitude), renal), endocrine or dismetabolic, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or pain condition, dermatological or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with scars or tattoos on the forearms, or with evidence of sunburn, or excessively hairy volar forearms.
* History of febrile illness within 5 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Mean blood perfusion (calculated as area under the effect curve [AUEC]) between 40 and 60 minutes post administration of capsaicin in the 3 cm x 3 cm area of capsaicin application. | 1 day

SECONDARY OUTCOMES:
Mean blood perfusion (calculated as AUEC), between 40 and 60 minutes post administration of capsaicin in the 12 cm x 5 cm area of laser Doppler scanning. | 1 day
Peak blood flow perfusion following the first use of the Peltier device between 0 and 30 minutes following termination of heat application in the 3 cm x 3 cm area of capsaicin application. | 1 day
Peak blood flow perfusion following the first use of the Peltier device between 0 and 30 minutes following termination of heat application in the 12 cm x 5 cm area of laser Doppler scanning. | 1 day
Peak blood flow perfusion following the second use of the Peltier device between 0 and 30 minutes following termination of heat application in the 3 cm x 3 cm area of capsaicin application. | 1 day
Peak blood flow perfusion following the second use of the Peltier device between 0 and 30 minutes following termination of heat application in the 12 cm x 5 cm area of laser Doppler scanning. | 1 day
Mean blood perfusion (calculated as AUEC) post first use of the Peltier device between 0 and 30 minutes following termination of heat application in the 3 cm x 3 cm area of capsaicin application. | 1 day
Mean blood perfusion (calculated as AUEC) post first use of the Peltier device between 0 and 30 minutes following termination of heat application in the 12 cm x 5 cm area of capsaicin application. | 1 day
Mean blood perfusion (calculated as AUEC) post second use of the Peltier device between 0 and 30 minutes following termination of heat application in the 3 cm x 3 cm area of capsaicin application. | 1 day
Mean blood perfusion (calculated as AUEC) post second use of the Peltier device between 0 and 30 minutes following termination of heat application in the 12 cm x 5 cm area of capsaicin application. | 1 day
Pain Intensity Scores as measured by an 11 point Numerical Rating Scale (NRS) 30-60 minutes post topical application of capsaicin cream. | 1 day
Pain Intensity Scores as measured by an 11 point Numerical Rating Scale (NRS) immediately following the first and second application of the heat stimulus. | 1 day
Plasma level of PF 06305591. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5281005&StudyName=Effect%20Of%20PF-06305591%20On%20Capsaicin%20And%20Capsaicin/Heat-Induced%20Neurogenic%20Flare